CLINICAL TRIAL: NCT01185288
Title: A Multicenter, Double-Blind, Randomized, Parallel-Arm Study to Determine the Effect of Methotrexate Dose on Clinical Outcome and Ultrasonographic Signs in Subjects With Moderately to Severely Active Rheumatoid Arthritis Treated With Adalimumab (MUSICA)
Brief Title: A Study to Determine the Effect of Methotrexate (MTX) Dose on Clinical Outcome and Ultrasonographic Signs in Subjects With Moderately to Severely Active Rheumatoid Arthritis (RA) Treated With Adalimumab (MUSICA)
Acronym: MUSICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-071
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab + Low Dose Methotrexate (Experimental): Open-label adalimumab (40 mg subcutaneous every other week) plus blinded, low dose methotrexate (7.5 mg orally once weekly).
  Interventions: Biological: Adalimumab; Drug: Methotrexate
- Adalimumab + High Dose Methotrexate (Active Comparator): Open-label adalimumab (40 mg subcutaneous every other week) plus blinded, high dose methotrexate (20 mg orally once weekly).
  Interventions: Biological: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Biological: Adalimumab — Adalimumab in pre-filled syringes
  Other Names: ABT-D2E7; Humira
Drug: Methotrexate — Methotrexate capsule

SUMMARY:
This study will investigate the efficacy of both low and high doses of methotrexate (MTX) in combination with open-label adalimumab (ADA) in patients who have had an inadequate response to high dose of MTX. The study will also evaluate the pharmacokinetics and safety of the two regimens of MTX in combination with ADA in participants with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with moderately to severely active rheumatoid arthritis
* Subjects must have a DAS28(CRP) (Disease Activity Score using C-Reactive Protein) greater than or equal to 3.2 at baseline (there is no minimum CRP score required to qualify)
* Subjects must have at least 5/68 tender joints plus 5/66 swollen joints assessed at screening or baseline
* Subject must treated with and MTX (methotrexate) dose (oral and/or injectable) of 15 mg or more per week (no upper limit on dose) for at least 12 weeks prior to screening
* Subject is either biologic-naïve or has only one prior biologic disease-modifying antirheumatic drug (i.e. abatacept, anakinra, certolizumab, etanercept, golimumab, infliximab, or tocilizumab)

Exclusion Criteria:

* Previous exposure to adalimumab (Humira), rituximab (Rituxan), natalizumab (Tysabri), efalizumab (Raptiva)
* Subject has been treated with intra-articular or parenteral administration of corticosteroids within 4 weeks of screening
* Subject has diagnosis or history of gout or pseudogout
* Subject has undergone joint surgery within 12 weeks of screening (at joints to be assessed by ultrasound)
* Subject has history of chronic arthritis diagnosed before age 16 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Carlson, MD, Study Director — AbbVie
Locations (49):
- United States (46):
  - Site Reference ID/Investigator# 38982, Huntsville, Alabama
  - Site Reference ID/Investigator# 38686, Tuscaloosa, Alabama
  - Site Reference ID/Investigator# 42044, Mesa, Arizona
  - Site Reference ID/Investigator# 37983, Phoenix, Arizona
  - Site Reference ID/Investigator# 44823, Little Rock, Arkansas
  - Site Reference ID/Investigator# 37981, Hemet, California
  - Site Reference ID/Investigator# 40208, Long Beach, California
  - Site Reference ID/Investigator# 38423, Sacramento, California
  - Site Reference ID/Investigator# 38204, Victorville, California
  - Site Reference ID/Investigator# 40762, Walnut Creek, California
  - Site Reference ID/Investigator# 43049, Danbury, Connecticut
  - Site Reference ID/Investigator# 38687, Jacksonville, Florida
  - Site Reference ID/Investigator# 40105, Miami, Florida
  - Site Reference ID/Investigator# 38083, Sarasota, Florida
  - Site Reference ID/Investigator# 38688, Lawrenceville, Georgia
  - Site Reference ID/Investigator# 38689, Meridian, Idaho
  - Site Reference ID/Investigator# 38085, Rock Island, Illinois
  - Site Reference ID/Investigator# 40128, Springfield, Illinois
  - Site Reference ID/Investigator# 38981, Bowling Green, Kentucky
  - Site Reference ID/Investigator# 38086, Covington, Louisiana
  - Site Reference ID/Investigator# 40125, Fall River, Massachusetts
  - Site Reference ID/Investigator# 65490, Las Vegas, Nevada
  - Site Reference ID/Investigator# 40124, Clifton, New Jersey
  - Site Reference ID/Investigator# 38978, Freehold, New Jersey
  - Site Reference ID/Investigator# 40123, Voorhees Township, New Jersey
  - Site Reference ID/Investigator# 38264, Smithtown, New York
  - Site Reference ID/Investigator# 38983, The Bronx, New York
  - Site Reference ID/Investigator# 38263, Asheville, North Carolina
  - Site Reference ID/Investigator# 38261, Greenville, North Carolina
  - Site Reference ID/Investigator# 39024, Mayfield Village, Ohio
  - Site Reference ID/Investigator# 40127, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 38202, Bend, Oregon
  - Site Reference ID/Investigator# 39023, Eugene, Oregon
  - Site Reference ID/Investigator# 38265, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 38082, Jackson, Tennessee
  - Site Reference ID/Investigator# 37980, Dallas, Texas
  - Site Reference ID/Investigator# 44888, Dallas, Texas
  - Site Reference ID/Investigator# 43050, Houston, Texas
  - Site Reference ID/Investigator# 43735, San Antonio, Texas
  - Site Reference ID/Investigator# 44344, Richmond, Virginia
  - Site Reference ID/Investigator# 40210, Seattle, Washington
  - Site Reference ID/Investigator# 38084, Seattle, Washington
  - Site Reference ID/Investigator# 38542, Seattle, Washington
  - Site Reference ID/Investigator# 38424, Spokane, Washington
  - Site Reference ID/Investigator# 38203, Tacoma, Washington
  - Site Reference ID/Investigator# 38087, Franklin, Wisconsin
- Puerto Rico (3):
  - Site Reference ID/Investigator# 60850, San Juan
  - Site Reference ID/Investigator# 38691, San Juan
  - Site Reference ID/Investigator# 60851, Vega Baja

REFERENCES:
- [Derived] Kaeley GS, MacCarter DK, Pangan AL, Wang X, Kalabic J, Ranganath VK. Clinical Responses and Synovial Vascularity in Obese Rheumatoid Arthritis Patients Treated with Adalimumab and Methotrexate. J Rheumatol. 2018 Dec;45(12):1628-1635. doi: 10.3899/jrheum.171232. Epub 2018 Sep 1. PMID 30173153
- [Derived] Kaeley GS, MacCarter DK, Goyal JR, Liu S, Chen K, Griffith J, Kupper H, Garg V, Kalabic J. Similar Improvements in Patient-Reported Outcomes Among Rheumatoid Arthritis Patients Treated with Two Different Doses of Methotrexate in Combination with Adalimumab: Results From the MUSICA Trial. Rheumatol Ther. 2018 Jun;5(1):123-134. doi: 10.1007/s40744-018-0105-7. Epub 2018 Mar 24. PMID 29574622
- [Derived] Burmester GR, Kaeley GS, Kavanaugh AF, Gabay C, MacCarter DK, Nash P, Takeuchi T, Goss SL, Rodila R, Chen K, Kupper H, Kalabic J. Treatment efficacy and methotrexate-related toxicity in patients with rheumatoid arthritis receiving methotrexate in combination with adalimumab. RMD Open. 2017 Sep 17;3(2):e000465. doi: 10.1136/rmdopen-2017-000465. eCollection 2017. PMID 28955494
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Kaeley GS, Evangelisto AM, Nishio MJ, Goss SL, Liu S, Kalabic J, Kupper H. Methotrexate Dosage Reduction Upon Adalimumab Initiation: Clinical and Ultrasonographic Outcomes from the Randomized Noninferiority MUSICA Trial. J Rheumatol. 2016 Aug;43(8):1480-9. doi: 10.3899/jrheum.151009. Epub 2016 Jun 15. PMID 27307526
- [Derived] Kaeley GS, Nishio MJ, Goyal JR, MacCarter DK, Wells AF, Chen S, Kupper H, Kalabic J. Changes in Ultrasonographic Vascularity Upon Initiation of Adalimumab Combination Therapy in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate. Arthritis Rheumatol. 2016 Nov;68(11):2584-2592. doi: 10.1002/art.39751. Epub 2016 Sep 29. PMID 27214046
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Started | 154 | 155
Completed | 135 | 139
Not Completed | 19 | 16
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 2 | 5
Not completed — Lack of Efficacy | 2 | 0
Not completed — Investigator discretion | 1 | 0
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate | Total
Number analyzed (Participants) | 154 | 155 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.11) | 54.5 (11.09) | 54.8 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 111 | 231
  Male | 34 | 44 | 78

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score for 28 Joints Based on C-reactive Protein (DAS28[CRP]) at Week 24
Description: The DAS28(CRP) score includes 28 tender joint counts, 28 swollen joint counts, C-reactive protein, and participant's global assessment of disease activity. Scores on the DAS28(CRP) range from 0 to 10. A DAS28(CRP) score ≥ 5.1 indicates high disease activity, and a DAS28(CRP) score < 2.6 indicates clinical remission. Least squares means and 95% CI were from 2-way ANCOVA model with effects for baseline DAS28(CRP) value, treatment group, and prior methotrexate dose group.
Time Frame: Week 24
Population: All participants who were randomized and received at least one dose of study medication (intent to treat). Missing responses were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
scores on a scale | 4.11 [3.88 to 4.34] | 3.75 [3.52 to 3.97]

2. Secondary Outcome: Percentage of Participants With Power Doppler Ultrasound (PD U/S) Score for Synovial Vascularity Improvement by 30% at Week 24
Description: PD U/S assessed the severity of synovial inflammation in both hands (bilateral wrists, metacarpophalangeal joints 2, 3, 5, and metatarsophalangeal joint 5). Bilateral images based on dorsal midline imaging of the wrist, dorsal and volar imaging of metacarpophalangeal joints, and dorsal imaging alone of metatarsophalangeal joints are scored using a 4-grade scale: grade 0 or normal = normal joint (no Doppler signal); grade 1 or mild = mild synovitis (≤ 3 isolated signals); grade 2 or moderate = moderate synovitis (> 3 isolated signals or a confluent signal in < 50% of synovial area); grade 3 or marked = marked synovitis (signals in ≥ 50% of the synovial area). Each image is rated 0 to 3, for a total possible score ranging from 0 to 48 (16*0, 16*3) for 2 hands. Higher grade/score=more severe disease. Change = week 24 score - baseline score.
Time Frame: Baseline, 24 weeks
Population: All participants who were randomized and received at least one dose of study medication (intent to treat). Missing responses were imputed by carrying forward the value at early termination visit (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
percentage of participants | 45.45 | 52.38

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% (ACR50) Criteria Response at Week 24
Description: Response, as defined by ACR50 criteria at week 24. A participant is a responder if the following 3 criteria for improvement from baseline are met: ≥ 50% improvement in tender joint count; ≥ 50% improvement in swollen joint count; and ≥ 50% improvement in at least 3 of the 5 following parameters: physician global assessment of disease activity, participant global assessment of disease activity, participant assessment of pain, disability index of the health assessment questionnaire, and acute phase reactant value (C-reactive protein).
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
percentage of participants | 29.80 | 37.66

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% (ACR70) Criteria Response at Week 24
Description: Response, as defined by ACR70 criteria at week 24. A participant is a responder if the following 3 criteria for improvement from baseline are met: ≥ 70% improvement in tender joint count; ≥ 70% improvement in swollen joint count; and ≥ 70% improvement in at least 3 of the 5 following parameters: physician global assessment of disease activity, participant global assessment of disease activity, participant assessment of pain, disability index of the health assessment questionnaire, and acute phase reactant value (C-reactive protein).
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
percentage of participants | 13.25 | 20.13

5. Secondary Outcome: Percentage of Participants With a Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) ≤ -0.22 at Week 24
Description: The HAQ-DI is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0), with some difficulty (1), with much difficulty (2), and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (no disability) to 3 (very severe, high dependency disability). The minimal clinically important difference (MCID) defined for the HAQ-DI is a change from baseline of ≤ -0.22. Normal physical function is defined by HAQ-DI score of < 0.5. Negative change from baseline in the overall score indicates improvement.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
percentage of participants | 63.58 | 65.58

6. Secondary Outcome: Percent Change From Baseline in Medical Outcomes Study Version II (MOS) Sleep Problem Index 9 at Week 24
Description: The least squares mean percentage change in MOS Sleep Problem Index 9 from baseline to week 24. The MOS Sleep Problem Index 9 consists of 9 questions to assess sleep, including how long it takes the participant to fall asleep (1=0 to 15 minutes, to 5=more than 60 minutes); and aspects of related to quality of sleep, including how often the participant felt that the sleep was not quiet, felt rested upon waking, awakened short of breath or with a headache, felt drowsy during the day, had trouble falling sleep, how often were awaken, had trouble staying awake during the day, and got needed amount of sleep (1=all the time; 5=none of the time). Least squares means and 95% CI were from 2-way ANCOVA model with effects for baseline MOS Sleep Problem Index value, treatment group, and prior methotrexate dose group.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
percent change | -15.42 [-25.36 to -5.49] | -17.27 [-27.95 to -7.58]

7. Other Pre Specified Outcome: Serum Adalimumab Trough Concentrations at Week 24
Description: Serum trough concentrations of adalimumab assessed at week 24 (24 weeks after the 1st dose).
Time Frame: Week 24
Population: All participants with available pharmacokinetics at week 24: For Adalimumab + Low Dose Methotrexate, n = 134; for Adalimumab + High Dose Methotrexate, n = 140.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Number analyzed (Participants) | 154 | 155
µg/mL | 7.1 (6.2) | 8.6 (5.2)

ADVERSE EVENTS:
Time Frame: AEs that occurred from the time of study drug administration until 70 days after last dose (total 34 weeks). SAEs were to be collected from the time that informed consent was obtained until 70 days after last dose (total 41 weeks).
Arm/Group | Adalimumab + Low Dose Methotrexate | Adalimumab + High Dose Methotrexate
Serious Adverse Events (participants affected / at risk) | 6/154 | 11/155
Other Adverse Events (participants affected / at risk) | 57/154 | 48/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Low Dose Methotrexate (N=154) | Adalimumab + High Dose Methotrexate (N=155)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
ABSCESS SOFT TISSUE (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 1
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Low Dose Methotrexate (N=154) | Adalimumab + High Dose Methotrexate (N=155)
DIARRHOEA (Gastrointestinal disorders) | 9 | 6
NAUSEA (Gastrointestinal disorders) | 15 | 16
FATIGUE (General disorders) | 14 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 | 12
URINARY TRACT INFECTION (Infections and infestations) | 8 | 11
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 9 | 5
DIZZINESS (Nervous system disorders) | 10 | 9
HEADACHE (Nervous system disorders) | 10 | 9
ALOPECIA (Skin and subcutaneous tissue disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.